CLINICAL TRIAL: NCT01592539
Title: Skin Blood Flow in Patients With Type 1 Diabetes Mellitus Compared to Normal Controls
Status: Completed | Type: Observational
Sponsor: Creighton University (Other)
Responsible Party: Principal Investigator, Laura Armas, Assistant Professor, Creighton University
Other Study IDs: Creighton11
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Type 1 Diabetes,; Bone
Keywords: Type 1 Diabetes; Bone
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case: Patients with Type 1 Diabetes Mellitus
- Control: Age and sex matched healthy controls.

SUMMARY:
The effects of high serum glucose on bone could be direct or could be indirect through its effects on the microvasculature. Previous studies by Rendell et al and Brugler et al have found significant differences in skin blood flow between diabetics and control. The investigators are proposing that blood flow measurements of the skin may be correlated with bone remodeling rates in iliac bone biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Must have completed a previous study.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with Type 1 DM
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2012-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura AG Armas, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States